CLINICAL TRIAL: NCT01032005
Title: Double Fortified Salt Intervention and Work Performance (Productivity) of Women Plantation Workers in West Bengal, India
Brief Title: Efficacy of Double Fortified Salt (DFS) to Improve Work Productivity in Women in India
Acronym: DFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Micronutrient Initiative (Other)
Collaborators: McGill University (Other); Cornell University (Other); The Mathile Institute for the Advancement of Human Nutrition (Other)
Responsible Party: Dr. Grace Marquis, McGill University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DFS efficacy trial
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Anemia; Iron Deficiency
MeSH Terms: conditions — Anemia; Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fortified salt (Placebo Comparator): Common table salt that has been fortified with iodine only
  Interventions: Other: double fortified salt
- Double fortified salt (Experimental): Common table salt that has been fortified with iron and well as the usual iodine
  Interventions: Other: double fortified salt

INTERVENTIONS:
Other: double fortified salt — Refined salt of particle size < 1 mm iodized with potassium iodate (KIO3) at a concentration of 30 µg I/g salt at the factory will be purchased and blended with encapsulated Ferrous Fumarate premix containing 15% iron. Premix to salt ratio of 1 to 150 will be used to arrive at 1000 ppm elemental iron in the final product.

SUMMARY:
The main objective of the present study is to assess the impact of double fortified salt containing iron and iodine on work performance (productivity) of women plantation workers in India. Efficacy studies have shown that salt double-fortified with iodine and iron can significantly reduce the incidence rates of iron-deficiency anemia (IDA) and iodine-deficiency disorders. Double-fortified salt (DFS) can be prepared by mixing microencapsulated iron compounds into conventionally iodated salt (Yuan et al, 2008). Iron deficiency anemia affects the work productivity and physical activity. Many studies have shown that when the individuals with low Hb received iron supplement, their work performance improved markedly. Animal studies have demonstrated that iron deficient anemic rats had a lower work tolerance as measured by oxygen consumption than the adult rats with normal Hb levels (Ohira et al, 1981). Several human studies have demonstrated the effect of iron supplementation on endurance capacity and work productivity in women (Zhu and Haas, 1997, 1998; Edgerton et al., 1979). Many human studies have also examined the possible linkages between iron deficiency and concurrent cognitive or behavioral outcomes. Iron supplementation effective in reducing iron-deficiency anemia would also result in better behavioral and developmental outcome. Many studies found that IDA had a great influence on cognitive functions in infants and school children (Lozoff et al., 2003, 1998 and Friel et al., 2003). However, studies of IDA and cognitive function in adults are few and controversial.

This study will assess iron status and physical and mental performance at 2 time points, before and after approximately 10 months during which a controlled intervention will take place on tea estates at the Panighatta Tea Garden near Siliguri, West Bengal. Subjects will be women between 18 and 50 years of age who are actively employed as full time tea pickers. The study requires that 2 experimental groups of subjects be identified: a) an experimental group that consumes double fortified salt (DFS) containing iron + iodine, and b) a control group that consumes only iodized salt (IS).

ELIGIBILITY:
Inclusion Criteria:

* Experienced, permanent, full-time tea pickers who plan to work for at least 2 picking seasons

Exclusion Criteria:

* Pregnant and lactating women
* Women with physical or mental disabilities that inhibit their ability to understand the study procedures or conduct their usual work (tea picking)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 248 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Work productivity (daily weight of tae picked) | endline (after 10 mo consumption of DFS)

SECONDARY OUTCOMES:
Anemia and iron status | Endline (after 10 mo consumption of DFS)
Cognitive function | Endline after 10 mo consumption of DFS

CONTACTS AND LOCATIONS:
Overall Officials: Grace Marquis, PhD, Principal Investigator — McGill University
Locations (1):
- Micronutrient Initiative, Panighatta Tea Estate, West Bengal, India

REFERENCES:
- [Background] Andersson M, Thankachan P, Muthayya S, Goud RB, Kurpad AV, Hurrell RF, Zimmermann MB. Dual fortification of salt with iodine and iron: a randomized, double-blind, controlled trial of micronized ferric pyrophosphate and encapsulated ferrous fumarate in southern India. Am J Clin Nutr. 2008 Nov;88(5):1378-87. doi: 10.3945/ajcn.2008.26149. PMID 18996875
- [Background] Edgerton VR, Gardner GW, Ohira Y, Gunawardena KA, Senewiratne B. Iron-deficiency anaemia and its effect on worker productivity and activity patterns. Br Med J. 1979 Dec 15;2(6204):1546-9. doi: 10.1136/bmj.2.6204.1546. PMID 534861
- [Background] Haas JD, Brownlie T 4th. Iron deficiency and reduced work capacity: a critical review of the research to determine a causal relationship. J Nutr. 2001 Feb;131(2S-2):676S-688S; discussion 688S-690S. doi: 10.1093/jn/131.2.676S. PMID 11160598
- [Background] Vinodkumar M, Rajagopalan S, Bhagwat IP, Singh S, Parmar BS, Mishra OP, Upadhyay SS, Bhalia NB, Deshpande SR. A multicenter community study on the efficacy of double-fortified salt. Food Nutr Bull. 2007 Mar;28(1):100-8. doi: 10.1177/156482650702800111. PMID 17718017
- [Derived] Nevins JE, Venkatramanan S, Mehta S, Haas JD. Predicting potential to benefit from an iron intervention: a randomized controlled trial of double-fortified salt in female Indian tea pluckers. Public Health Nutr. 2019 Dec;22(18):3416-3425. doi: 10.1017/S1368980019001800. Epub 2019 Jul 25. PMID 31342886
- [Derived] Wenger MJ, Murray-Kolb LE, Nevins JE, Venkatramanan S, Reinhart GA, Wesley A, Haas JD. Consumption of a Double-Fortified Salt Affects Perceptual, Attentional, and Mnemonic Functioning in Women in a Randomized Controlled Trial in India. J Nutr. 2017 Dec;147(12):2297-2308. doi: 10.3945/jn.117.251587. Epub 2017 Oct 11. PMID 29021371
- [Derived] Haas JD, Rahn M, Venkatramanan S, Marquis GS, Wenger MJ, Murray-Kolb LE, Wesley AS, Reinhart GA. Double-fortified salt is efficacious in improving indicators of iron deficiency in female Indian tea pickers. J Nutr. 2014 Jun;144(6):957-64. doi: 10.3945/jn.113.183228. Epub 2014 Apr 17. PMID 24744318